CLINICAL TRIAL: NCT07217496
Title: Phase Ib Trial Combining N-803 and Pembrolizumab With Shorter Duration of Enfortumab Vedotin in Treatment-Naïve Patients With Metastatic Urothelial Carcinoma
Brief Title: N-803 in Combination With Pembrolizumab and Enfortumab Vedotin for Treatment of Urothelial Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vadim S Koshkin (Other)
Collaborators: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Vadim S Koshkin, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25525; NCI-2025-07330 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Urothelial Carcinoma; Urothelial Carcinoma; Locally Advanced Urothelial Carcinoma; Urothelial Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — ALT-803; enfortumab vedotin; pembrolizumab; Phantoms, Imaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (EV, N-803, pembrolizumab) (Experimental): Participants with unresectable locally advanced (LA) or metastatic urothelial carcinoma (mUC) will receive N-803 plus Enfortumab Vedotin (EV) and Pembrolizumab on Day 1 and EV on Day 8 in a repeated 3-week cycle until disease progression or unacceptable toxicity. EV treatment is provided up to 12 cycles. Participants with confirmed clinical benefit based on Response Evaluation Criteria in Solid Tumors (RECIST v1.1) at the second or third scan (between 8 to 12 cycles on treatment) will discontinue EV treatment at investigator discretion. After participants discontinue EV treatment, participants may continue to receive N-803 and Pembrolizumab treatment up to 2 years.
  Interventions: Drug: Nogapendekin Alfa Inbakicept (N803); Drug: Enfortumab Vedotin (EV); Drug: Pembrolizumab; Procedure: Research Biospecimen Collection; Procedure: Radiographic Imaging; Procedure: Tumor Biopsy

INTERVENTIONS:
Drug: Nogapendekin Alfa Inbakicept (N803) — Given subcutaneously (SC)
  Other Names: Nogapendekin Alfa Inbakicept; N803
Drug: Enfortumab Vedotin (EV) — Given intravenously (IV)
  Other Names: Enfortumab Vedotin
Drug: Pembrolizumab — Given intravenously (IV)
  Other Names: Keytruda
Procedure: Research Biospecimen Collection — Undergo blood collection for research purposes
Procedure: Radiographic Imaging — Undergo radiographic imaging for disease assessment
  Other Names: Magnetic Resonance Imaging (MRI); Computed tomography (CT)
Procedure: Tumor Biopsy — Undergo tumor biopsy

SUMMARY:
This phase Ib trial will investigate the effect of N-803 in combination with pembrolizumab and enfortumab vedotin in treating participants with urothelial cancer that has spread to nearby tissue or lymph nodes (locally advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and tolerability of the treatment regimen (N-803, enfortumab vedotin, and pembrolizumab).

II. To assess 12-month progression-free survival (PFS) of participants with locally advanced or metastatic urothelial carcinoma (mUC) receiving enfortumab vedotin (EV) plus pembrolizumab and N-803.

SECONDARY OBJECTIVE:

I. To evaluate the preliminary efficacy of the treatment regimen (EV, pembrolizumab, and N-803) as measured by complete response rate (CRR), objective response rate (ORR), clinical benefit rate (CBR), 12-month overall survival (12-OS), median duration of response (mDOR), median progression-free survival (mPFS) and median overall survival (mOS).

EXPLORATORY OBJECTIVES:

I. To determine the immune status of the tumor microenvironment using multiplex immunohistochemistry (IHC) and identify potential correlations with participant outcomes.

II. To determine T-cell receptor (TCR) clonality.

III. To analyze tumor/immune gene expression profiles, DNA methylation, DNA damage response and repair (DDR) genes [e.g., BRCA1/2, ERCC1/2]).

IV. Observe changes in circulating tumor DNA (ctDNA).

V. To monitor the maintenance of absolute lymphocyte counts (ALC) relative to baseline, throughout the course of treatment.

OUTLINE:

This is an open-label, single center, phase Ib single-arm trial with a safety lead-in cohort. Participants will receive treatment for up to 12 cycles administered. Depending on response, participants may continue treatment with pembrolizumab and N-803 for maximum of 2 years. Participants will undergo safety follow-up approximately 30 days following the end of study treatment and be followed for survival until death (any cause) or end of study for a up to 5 years from start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically confirmed locally advanced (LA)/ metastatic urothelial carcinoma (mUC), including UC originating from the renal pelvis, ureters, bladder, or urethra. Mixed-cell type tumors are eligible as long as > 50% urothelial component is present (mixed histology other than small cell/ neuroendocrine are allowed).
3. No prior systemic treatment for LA/mUC.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) <= 2.
5. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.
6. Prior perioperative systemic therapy including neoadjuvant or adjuvant chemotherapy, immune checkpoint inhibitors, and EV is allowed if treatment was completed > 12 months before trial enrollment.
7. Participants enrolling in the trial must agree with discontinuing EV upon demonstrating confirmed CR/PR/SD at the second or third scan timepoint on treatment (after 5.5 to 8 months of intended EV treatment).
8. Leukocytes ≥ 3,000/microliter (uL).
9. Absolute neutrophil count (ANC) ≥ 1,500/uL.
10. Platelets ≥ 100,000/uL.
11. Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (if previously abnormal due to non-malignant causes such as Gilbert's disease bilirubin ≤ 2 x ULN will be permitted.)
12. Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase (SGOT))/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal (ULN).
13. Creatinine clearance ≥ 30 mL/min/1.73 m^2 calculated using the Cockcroft-Gault equation.
14. Must have archival tumor tissue available or have disease amenable to a fresh biopsy for diagnosis confirmation and correlative studies.
15. Human immunodeficiency virus (HIV)-infected individuals with undetectable viral load within 6 months are eligible for this trial. Trial participants who are on antiretroviral therapy (ART) should be on established ART for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment.
16. For participants with history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable and the participant should be on suppressive antiviral therapy, if indicated. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured, with HCV viral load below the level of quantification. A participant who is HCV antibody (Ab) positive but HCV ribonucleic acid (RNA) negative due to prior treatment or natural resolution is eligible for this trial. For individuals with HCV infection who are currently on treatment, they are eligible if HCV viral load below the level of quantification. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
17. participants who are on beta blockers can enroll in the trial, but discontinuation of beta-blockers should be strongly considered at the time of initiating N-803. Beta blocker use can continue per physician discretion if necessary.

    * Note: Beta-blockers or other antihypertensives may be resumed on treatment when clinically indicated.
18. Agreement to practice effective contraception for female participants of child-bearing potential and non-sterile males. Female participants of child-bearing potential must agree to use effective contraception for up to 4 months after completion of therapy, and non-sterile male participants must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (e.g., vasectomy, tubal ligation), oral and injectable contraceptives, 2 forms of barrier methods (e.g., condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and hormonal therapy. For male participants with a female partner of child-bearing potential, the female partner must also agree to use effective contraception for up to 4 months after therapy was completed.
19. Able to understand and provide a signed informed consent that fulfills the relevant institutional review board (IRB) or independent ethics committee (IEC) guidelines.

Exclusion Criteria:

1. Symptomatic or untreated central nervous system (CNS) metastases.

   * Note: Participants with previously treated brain or CNS metastases are eligible if the participant has recovered from any acute effects of surgery or radiotherapy and do not require steroids (prednisone equivalent ≥ 10 mg daily), and any whole brain radiation therapy or any stereotactic radiosurgery was completed at least 2 weeks prior to initiation of therapy.
2. Participants with a history of active autoimmune disease and on active management with immunosuppressive agents within the past 2 years
3. Participants with a history of interstitial lung disease
4. Participants with congestive heart failure (New York Heart Association class III or IV)
5. Participants on systemic intravenous or oral corticosteroid therapy (prednisone equivalent ≥ 10 mg daily) or other immunosuppressive agents such as azathioprine or cyclosporin A are excluded. For these participants, these excluded treatments must be discontinued at least 1 week prior to enrollment for recent short course use (≤ 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (> 14 days).

   * Note: The use of corticosteroids as premedication for contrast-enhanced studies is allowed prior to enrollment and on study. participants requiring hormone replacement with corticosteroids if the steroids are administered only for the purpose of hormonal replacement or participants treated at doses ≤ 10 mg of prednisone or equivalent per day are allowed.
6. History of uncontrolled diabetes mellitus defined as hemoglobin A1c (HbA1c) ≥ 8%.
7. Grade ≥ 2 peripheral neuropathy at baseline.
8. Radiotherapy or major surgery within 2 weeks prior to treatment start.
9. History of another significant life-limiting malignancy within 2 years prior to the first dose of study drug. Participants with non-melanoma skin cancer, curatively treated localized prostate cancer, or carcinoma in situ of any type (if complete resection was done) are allowed.
10. History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to EV and/or pembrolizumab and/or N-803.
11. Participants who have received hematopoietic stem cell transplantation or solid organ transplantation.
12. Known active keratitis or corneal ulcerations.
13. Received or will receive a live vaccine within 30 days prior to the first administration of study intervention.

    * Note: Seasonal flu vaccines that do not contain a live virus are permitted. Locally approved Coronavirus disease of 2019 (COVID-19) vaccines are permitted.
14. Pregnant and nursing women.
15. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.
16. Severe uncontrolled intercurrent illness that would limit compliance with study requirements in the judgement of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with reported Treatment-Emergent Adverse Events | Up to 2 years
  Treatment emergent adverse events will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events version (v) 5.0.
Number of participants with reported Dose-limiting toxicities (DLTs) | Up to 28 days
  Safety will be evaluated by assessing for DLTs in the first 6 participants treated with the study drug combination. If >33% or >2 of the first six participants experiences a DLT, the dose will be reviewed, and study will be considered for modification.
Percentage of participants alive and progression free at 12 months (PFS12) | 12 months
  The percentage of participants alive and progression free at 12 months is defined from the date of first dose of study drugs (C1D1) to the date of disease progression or death (any cause), whichever occurs first, by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. If disease progression or death from any cause is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the PFS will be censored as the last available disease assessment. Kaplan Meier analyses will be used to estimate 12 month PFS with 90% confidence interval.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | Up to 2 years
  Defined as the portion of participants who experience a confirmed complete response (CR) per RECIST 1.1. Data will be collected from enrollment until the participant experiences disease progression, initiates subsequent anti-cancer therapy, or completes study participation (whichever occurs first).
Clinical Benefit Rate (CBR) | Up to 24 weeks
  Clinical benefit rate is defined as the proportion of participants who experience clinical benefit (CR, partial response (PR) or stable disease (SD)) for at least 24 weeks (two consecutive scans) per RECIST 1.1. criteria.
Objective Response Rate (ORR) | Up to 2 years
  Defined as the portion of participants who experience an objective response (confirmed complete response (CR) or confirmed partial response (PR)) per RECIST 1.1. ORR data will be collected from enrollment until the response has been confirmed, the participant experiences disease progression, initiates subsequent anti-cancer therapy, or completes study participation (whichever occurs first).
Median Overall Survival (OS) | Up to 5 years
  Defined as the amount of time that elapses between /the initiation of trial therapy (C1D1) and the time of death from any cause. OS data will be collected from enrollment until the participant completes study follow-up participation, experiences death from any cause or is documented as lost to follow up per institutional standard (whichever is sooner). If death from any cause is not observed prior to completing study participation, the OS will be censored as the time of the last available documentation of survival status. (Last available documentation of survival status is defined as the date of death or the latest of the following times: treatment discontinuation date, last dosing administration date, last disease assessment date, or the last follow up date when the participant was known to be alive.)
Median Duration of Response (DOR) | Up to 5 years
  Defined as the time that elapses between the first day of documented response to trial therapy and subsequent disease progression. For DOR analysis, response is defined as confirmed complete response (CR), or confirmed partial response (PR), per RECIST 1.1 and disease progression is defined as progressive disease (PD) per RECIST 1.1. If disease progression is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the DOR will be censored as the last available disease assessment.
Median Progression-Free Survival (PFS) | Up to 5 years
  Defined as the amount of time that elapses between the initiation of trial therapy (C1D1) and the day of first documented disease progression or death. If disease progression or death from any cause is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the PFS will be censored as the last available disease assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Vadim Koshkin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with study collaborators during the course of the study.
Supporting Information: Study Protocol, SAP